CLINICAL TRIAL: NCT04210804
Title: A Prophylactic Trial of Omega-3 Polyunsaturated Fatty Acids in Bipolar Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Brian Hallahan, Senior Lecturer, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12/12
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Bipolar Depression
Keywords: Omega-3; Bipolar Disorder; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: One month placebo run in prior to randomisation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 (Experimental): 1gEPA and 1gDHA in 200mls smoothie
  Interventions: Dietary Supplement: Smoothie 1g Eicosapentaneoic Acid (EPA) and 1g Docoshaexanoic Acid (DHA)
- Placebo (Placebo Comparator): 200mls smoothie without EPA or DHA. Looks and tastes identical to omega-3 arm
  Interventions: Dietary Supplement: Smoothie 1g Eicosapentaneoic Acid (EPA) and 1g Docoshaexanoic Acid (DHA)

INTERVENTIONS:
Dietary Supplement: Smoothie 1g Eicosapentaneoic Acid (EPA) and 1g Docoshaexanoic Acid (DHA) — 200mls Smoothie

SUMMARY:
This study is a 52 week double-blind placebo controlled study of omega-3 polyunsaturated fatty acids (PUFAs) in bipolar disorder (who have a history of 3 or more episodes) to ascertain if omega-3 PUFAs reduce the risk of further relapse for both / either depressive or (hypo)manic episodes.

This is a single-centre, 52 week, double-blind, randomised comparison of omega-3 PUFA (1g EPA and 1g DHA) versus placebo as adjunctive treatment in individuals with bipolar disorder

DETAILED DESCRIPTION:
Bipolar Disorder is a chronic disabling psychiatric disorder characterized by recurrent episodes of mania or hypomania and depression. Bipolar Disorder can be separated into bipolar I and bipolar II disorders with bipolar I disorder characterizing individuals who have episodes of mania and depression, and bipolar II disorder characterizing individuals who have episodes of depression with periods of hypomania, but not mania. Bipolar Disorder has an estimated prevalence of approximately 1% and a roughly equal gender ratio. Treatment of bipolar disorder is predominantly by pharmacological means with probably the most evidence still supporting the role of lithium both for the treatment of bipolar disorder and prophylaxis of further episodes (particularly (hypo)manic episodes.

A number of other standard mood stabiliser agents are often utilised including sodium valproate, carbamazepine and lamotrigine. Over the last 10 years, a number of antipsychotic agents have attained a licence for the treatment of bipolar disorder including olanzapine, quetiapine, asenapine and aripiprazole. All of these treatments are associated with significant adverse effects. For example, lithium has been associated with hypothyroidism and diabetes insipidus, interacts with a variety of other agents including non-steroidal anti-inflammatory drugs, diuretics and requires careful blood monitoring to ensure that the individuals blood level is within a therapeutic range (to avoid toxicity or subclinical treatment). Sodium Valproate is associated with several adverse effects; principal amongst these is teratogenesis in pregnancy, but also alopecia and a hand tremor. Carbamazepine is associated with blood dyscrasias and hyponatraemia and interacts with many medications. Lamotrigine has been utilised for the treatment of bipolar depression, however it can take several months of treatment before one reaches therapeutic doses, and severe skin rashes occasionally occur. In relation to the antipsychotic agents, olanzapine is associated with significant weight gain, somnolence and metabolic syndrome, quetiapine is associated with hypotension and somnolence, aripiprazole is associated with akathisia and asenapine is associated with dizziness and somnolence. Whilst psychotherapy has demonstrated some benefit for the treatment of bipolar depression, to date, the role of psychotherapy for the management of (hypo)mania remains limited.

The putative role of omega-3 polyunsaturated fatty acids (omega-3 PUFAs) principally eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in the treatment of mood disorders has been supported by a wide variety of epidemiological observations, tissue compositional comparisons, clinical and treatment studies. For example, cross-national studies have found a substantially higher incidence of depression, suicide, and bipolar disorder in cultures with low omega-3 PUFA intake (due to low levels of fish consumption) with low levels of fish consumption also independently associated with symptoms of depression. Lower concentrations of both EPA and DHA have been found in red blood cells of depressed individuals compared to healthy controls, and the ratio of EPA to the omega-6 PUFA arachidonic acid (AA) has been demonstrated both in depression and in mania. The most specific evidence for central tissue compositional deficits is the finding of lower DHA in the post-mortem orbitofrontal cortex of patients with both major depressive disorder and bipolar disorder.

Several randomised controlled trials have also demonstrated a benefit for omega-3 PUFAs in depression, although these findings are not universal and meta-analyses have noted substantial heterogeneity in these findings. Although there have been multiple treatment trials examining the putative antidepressant effect of omega-3 PUFAs in recurrent depressive disorder, we are aware of only six randomised double-blind placebo-controlled trials to date that have investigated if omega-3 PUFAs have a therapeutic role in bipolar disorder. In these trials, results have been contradictory with two studies demonstrating a benefit for omega-3 PUFAs compared to placebo, with both of these trials demonstrating a reduction in depressive but not manic symptoms. with one study using high dose EPA (6.2g) and DHA (3.4g) for a period of 16 weeks, and another using lower formulations of EPA alone at doses of 1g or 2g for a period of 12 weeks. In relation to the five negative trials to date; DHA alone (2g) was administered to a small cohort of euthymic bipolar individuals (n=10; 6 = DHA, 4 = placebo) over a 52 week period in one study. Another study administered high dose EPA (6g) however, the drop-out rate was high at 54%. Two trials administered alpha-linolenic acid (ALA) (the parent omega-3 PUFA) or a mixture of PUFAs (3g EPA and 2g DHA) and pyrimidine cytidine (n=15), with no benefit noted. One final study was presented in the form of a letter to the editor and conducted in a small cohort of 15 individuals with minimal data provided.

Therefore, it is unclear if omega-3 PUFAs have a therapeutic role in bipolar disorder. Studies to date have utilised a variety of PUFA formulations, for short time periods and have included either modest numbers or have had high drop-out rates.

Humans have limited capacity to synthesize EPA or DHA de novo and make only limited amounts of DHA from the dietary precursor omega-3, ALA. Fish and shellfish are the primary dietary sources of preformed EPA and DHA. Both of these omega-3 PUFAs play an important role in many physiological processes including inflammation, and DHA is selectively concentrated in synaptic neuronal membranes. EPA has significant immunological neurotrophic and hormone like activities which may explain to date, the greater evidence for its antidepressant efficacy. EPA is more rapidly incorporated into membrane phospholipids, increasing inflammation resolution of circulating mononuclear cells, resulting in attenuated production of the pro-inflammatory cytokines, interleukin-1 (IL-1) and tumor necrosis factor alpha (TNF). Both major depressive disorder (MDD) and bipolar disorder are associated with increased circulating pro-inflammatory cytokines including IL-1, IL-6 and TNF-α and perhaps the demonstrated antidepressant effects of EPA may be related in some part to its anti-inflammatory role. Other postulated mechanisms for a putative role of omega-3 PUFAs in bipolar disorder include suppression of neuronal signalling, second messenger generation, calcium channel and protein kinase C activity and kindling. Western diets are deficient in omega-3 PUFAs, largely due to relatively low seafood consumption and the food industry preference for corn and soy oils high in the short-chain omega-6 PUFA acid linoleic acid. However, omega-3 PUFAs are becoming an increasingly popular over-the-counter dietary supplement and are an appealing option for treatment of both physical and psychiatric illness, given the perception that they are a "natural" substance and that they possess a very benign adverse effect profile.

To date, despite moderate evidence for the efficacy of omega-3 PUFAs in recurrent depressive disorder (major depressive illness), little is known in relation to the possible efficacy of omega-3 PUFAs in bipolar disorder. As stated, studies to date in bipolar disorder have occurred in individuals with euthymia or mild depression and the maximum trial duration as mentioned above except for one study with only 10 participants has been 16 weeks. Participants in this study will be adults (aged 18 or older) recruited from the local mental health service, which include a specialised bipolar disorder clinic (n=40) and 12 other out-patient clinics per week, where approximately another 160 individuals with bipolar disorder attend. Approximately 130 individuals attending the service would satisfy criteria for study inclusion and it is envisaged based on previous research by Hallahan and colleagues in the same population, that 70% (n=91) would be willing to engage in this treatment trial. If insufficient numbers are available to participate from the local mental health service, significant links with adjoining HSE West services (within 1 hour of Galway) have been developed for research purposes over the last seven years and additional participants could be attained.

After a complete description of the study, written informed consent will be obtained from all participants and signed agreement will be obtained from their treating psychiatrist. Previous studies demonstrating a treatment effect in depression and both positive bipolar disorder studies have had EPA as the sole or principal omega-3 PUFA, and thus the investigators felt that it was important that EPA was a significant component of the PUFA formulation. Based on a recent hierarchical meta-analysis conducted at NUI Galway, it is clear that EPA has some clinical benefit for depression and DHA as the predominant component in a PUFA formulation has no significant clinical benefit, however when both compounds were present, the beneficial effect was at least as efficacious (marginally more efficacious but not to a statistical significant level) than where EPA was the sole PUFA agent. Furthermore, as DHA enrichment and turnover in the brain is slow (unlike EPA), with a half-life of approximately 2.5 years, it is not surprising that relatively short RCTs would not demonstrate a benefit with DHA.

Consequently individuals who consent to participate in this study will take either the active agent which is Omega-3 PUFA: Dose = 1g Eicosapentaenoic Acid (EPA) and 1g Docosahexaenoic Acid (DHA) taken po as a juice (200ml; Smartfish Nutrifriend 2000). Placebo will look and taste identical to the active compound.

Omega-3 PUFAs are freely available to attain in a variety of health shops, pharmacies and in some general retail shops also. Consequently they are not in any phase of development, however their benefit, long established for physical conditions such as arthritis has also been postulated for mood disorders and evidence for benefit has been attained in a number of randomised controlled trials and meta-analyses with no associated adverse consequences.

After a 1-3 month placebo run in time, participants will take the active or placebo agent for 12 months.

No medical regulatory board approval was required (HPRA in Ireland) as this is a nutrient rather than a medication.

Aims Primary: Undertake a 52 week single-centre, double-blind, placebo controlled study of omega-3 polyunsaturated fatty acids (PUFAs) in bipolar disorder (who have a history of 3 or more episodes) to ascertain if omega-3 PUFAs reduce the risk of further relapse for both / either depressive or (hypo)manic episodes.

Secondary: Ascertain if there is any difference from baseline mood scores for both elation and depression for omega-3 PUFAs compared to placebo. The investigators wish to ascertain what proportion of individuals drop out of the study from both groups.

Statistical analysis will be carried out utilising the Statistical Package for Social Sciences 24 (SPSS 24) or other statistical programmes as deemed necessary. Significance will be set at 0.05 and all tests will be two-tailed. Parametric data will be analysed using student t-tests or analysis of co-variance where appropriate and non-parametric data will be analysed using chi-squared test. A repeated analysis of variance (ANOVA) with baseline rating scores entered as co-variates will be used to compare changes in psychopathology over time in the two groups. Survivor analysis (Kaplan-Meier) will also be utilised in this study.

No analysis has been conducted to date and the code for placebo or active groups has not been broken.

Psychometric Instruments utilised include the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID), the Beck Depression Inventory (BDI), the Hamilton Depression Rating Scale (HDRS), the Young Mania Rating Scale (YMRS), the Global Assessment of Functioning (GAF) scale and Clinical Global Impression (CGI).

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent and comply with the study protocol.
2. An established diagnosis of bipolar disorder (either type I or II) and have had at least 3 previous episodes of illness within the previous 5 years or 2 episodes in the last 12 months.

To be eligible for inclusion, each subject must meet each of the inclusion criteria at Screening (Visit 1) and must continue to fulfil these criteria at Baseline (Visit 2).

Exclusion Criteria:

* Severity of their bipolar disorder is such that participation in a clinical trial is not appropriate because of the risk of imminent self-harm or psychiatric admission,
* A concurrent medical condition (intracranial brain lesion),
* Medication (steroids) that may be accounting for the mood episodes,
* Participant is taking omega-3 PUFA supplements at the time of study entry or in the previous 12 weeks
* Individuals who are participating in another study where they are receiving a different investigational agent during the course, or within the 12 week period prior to their inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Episodes of Depression or Elation | 15 months (duration of trial and 3 month follow-up)
  Documented episodes of depression or elation noted in clinical notes, or re-hospitalisation or treatment change secondary to episode of depression or elation

SECONDARY OUTCOMES:
Psychometric Measures of Depression or Elation | 15 months (duration of trial and 3 month follow-up)
  Change from baseline in psychometric instruments
Adverse Effects | 15 months (duration of trial and 3 month follow-up)
  Presence of adverse effects secondary to intervention or placebo
Continuation rate | 15 months (duration of trial and 3 month follow-up)
  Study engagement rates between intervention and placebo arms
Time to relapse of depression or elation | 15 months (duration of trial and 3 month follow-up)
  Time to relapse of depression or elation

CONTACTS AND LOCATIONS:
Locations (1):
- NUI Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No
No plan for data sharing

REFERENCES:
- [Background] Adams PB, Lawson S, Sanigorski A, Sinclair AJ. Arachidonic acid to eicosapentaenoic acid ratio in blood correlates positively with clinical symptoms of depression. Lipids. 1996 Mar;31 Suppl:S157-61. doi: 10.1007/BF02637069. PMID 8729112
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Belmaker RH. Bipolar disorder. N Engl J Med. 2004 Jul 29;351(5):476-86. doi: 10.1056/NEJMra035354. No abstract available. PMID 15282355
- [Background] Caughey GE, Mantzioris E, Gibson RA, Cleland LG, James MJ. The effect on human tumor necrosis factor alpha and interleukin 1 beta production of diets enriched in n-3 fatty acids from vegetable oil or fish oil. Am J Clin Nutr. 1996 Jan;63(1):116-22. doi: 10.1093/ajcn/63.1.116. PMID 8604658
- [Background] Cetin T, Guloksuz S, Cetin EA, Gazioglu SB, Deniz G, Oral ET, van Os J. Plasma concentrations of soluble cytokine receptors in euthymic bipolar patients with and without subsyndromal symptoms. BMC Psychiatry. 2012 Sep 26;12:158. doi: 10.1186/1471-244X-12-158. PMID 23013558
- [Background] Chiu CC, Huang SY, Chen CC, Su KP. Omega-3 fatty acids are more beneficial in the depressive phase than in the manic phase in patients with bipolar I disorder. J Clin Psychiatry. 2005 Dec;66(12):1613-4. doi: 10.4088/jcp.v66n1219b. No abstract available. PMID 16401167
- [Background] da Silva TM, Munhoz RP, Alvarez C, Naliwaiko K, Kiss A, Andreatini R, Ferraz AC. Depression in Parkinson's disease: a double-blind, randomized, placebo-controlled pilot study of omega-3 fatty-acid supplementation. J Affect Disord. 2008 Dec;111(2-3):351-9. doi: 10.1016/j.jad.2008.03.008. Epub 2008 May 15. PMID 18485485
- [Background] Frangou S, Lewis M, McCrone P. Efficacy of ethyl-eicosapentaenoic acid in bipolar depression: randomised double-blind placebo-controlled study. Br J Psychiatry. 2006 Jan;188:46-50. doi: 10.1192/bjp.188.1.46. PMID 16388069
- [Background] Gertsik L, Poland RE, Bresee C, Rapaport MH. Omega-3 fatty acid augmentation of citalopram treatment for patients with major depressive disorder. J Clin Psychopharmacol. 2012 Feb;32(1):61-4. doi: 10.1097/JCP.0b013e31823f3b5f. PMID 22198441
- [Background] Goyens PL, Spilker ME, Zock PL, Katan MB, Mensink RP. Compartmental modeling to quantify alpha-linolenic acid conversion after longer term intake of multiple tracer boluses. J Lipid Res. 2005 Jul;46(7):1474-83. doi: 10.1194/jlr.M400514-JLR200. Epub 2005 Apr 16. PMID 15834128
- [Background] Gracious BL, Chirieac MC, Costescu S, Finucane TL, Youngstrom EA, Hibbeln JR. Randomized, placebo-controlled trial of flax oil in pediatric bipolar disorder. Bipolar Disord. 2010 Mar;12(2):142-54. doi: 10.1111/j.1399-5618.2010.00799.x. PMID 20402707
- [Background] Hallahan B, Hibbeln JR, Davis JM, Garland MR. Omega-3 fatty acid supplementation in patients with recurrent self-harm. Single-centre double-blind randomised controlled trial. Br J Psychiatry. 2007 Feb;190:118-22. doi: 10.1192/bjp.bp.106.022707. PMID 17267927
- [Background] Hallahan B, Ryan T, Hibbeln JR, Murray IT, Glynn S, Ramsden CE, SanGiovanni JP, Davis JM. Efficacy of omega-3 highly unsaturated fatty acids in the treatment of depression. Br J Psychiatry. 2016 Sep;209(3):192-201. doi: 10.1192/bjp.bp.114.160242. Epub 2016 Apr 21. PMID 27103682
- [Background] Hibbeln JR. Fish consumption and major depression. Lancet. 1998 Apr 18;351(9110):1213. doi: 10.1016/S0140-6736(05)79168-6. No abstract available. PMID 9643729
- [Background] Hibbeln JR. Seafood consumption, the DHA content of mothers' milk and prevalence rates of postpartum depression: a cross-national, ecological analysis. J Affect Disord. 2002 May;69(1-3):15-29. doi: 10.1016/s0165-0327(01)00374-3. PMID 12103448
- [Background] Hibbeln JR, Nieminen LR, Blasbalg TL, Riggs JA, Lands WE. Healthy intakes of n-3 and n-6 fatty acids: estimations considering worldwide diversity. Am J Clin Nutr. 2006 Jun;83(6 Suppl):1483S-1493S. doi: 10.1093/ajcn/83.6.1483S. PMID 16841858
- [Background] Hope S, Dieset I, Agartz I, Steen NE, Ueland T, Melle I, Aukrust P, Andreassen OA. Affective symptoms are associated with markers of inflammation and immune activation in bipolar disorders but not in schizophrenia. J Psychiatr Res. 2011 Dec;45(12):1608-16. doi: 10.1016/j.jpsychires.2011.08.003. Epub 2011 Sep 1. PMID 21889167
- [Background] Keck PE Jr, Mintz J, McElroy SL, Freeman MP, Suppes T, Frye MA, Altshuler LL, Kupka R, Nolen WA, Leverich GS, Denicoff KD, Grunze H, Duan N, Post RM. Double-blind, randomized, placebo-controlled trials of ethyl-eicosapentanoate in the treatment of bipolar depression and rapid cycling bipolar disorder. Biol Psychiatry. 2006 Nov 1;60(9):1020-2. doi: 10.1016/j.biopsych.2006.03.056. Epub 2006 Jun 30. PMID 16814257
- [Background] Khairova RA, Machado-Vieira R, Du J, Manji HK. A potential role for pro-inflammatory cytokines in regulating synaptic plasticity in major depressive disorder. Int J Neuropsychopharmacol. 2009 May;12(4):561-78. doi: 10.1017/S1461145709009924. Epub 2009 Feb 19. PMID 19224657
- [Background] Kraguljac NV, Montori VM, Pavuluri M, Chai HS, Wilson BS, Unal SS. Efficacy of omega-3 fatty acids in mood disorders - a systematic review and metaanalysis. Psychopharmacol Bull. 2009;42(3):39-54. PMID 19752840
- [Background] Lesperance F, Frasure-Smith N, St-Andre E, Turecki G, Lesperance P, Wisniewski SR. The efficacy of omega-3 supplementation for major depression: a randomized controlled trial. J Clin Psychiatry. 2011 Aug;72(8):1054-62. doi: 10.4088/JCP.10m05966blu. Epub 2010 Jun 15. PMID 20584525
- [Background] Lin PY, Su KP. A meta-analytic review of double-blind, placebo-controlled trials of antidepressant efficacy of omega-3 fatty acids. J Clin Psychiatry. 2007 Jul;68(7):1056-61. doi: 10.4088/jcp.v68n0712. PMID 17685742
- [Background] Marangell LB, Martinez JM, Zboyan HA, Kertz B, Kim HF, Puryear LJ. A double-blind, placebo-controlled study of the omega-3 fatty acid docosahexaenoic acid in the treatment of major depression. Am J Psychiatry. 2003 May;160(5):996-8. doi: 10.1176/appi.ajp.160.5.996. PMID 12727707
- [Background] Marangell LB, Suppes T, Ketter TA, Dennehy EB, Zboyan H, Kertz B, Nierenberg A, Calabrese J, Wisniewski SR, Sachs G. Omega-3 fatty acids in bipolar disorder: clinical and research considerations. Prostaglandins Leukot Essent Fatty Acids. 2006 Oct-Nov;75(4-5):315-21. doi: 10.1016/j.plefa.2006.07.008. Epub 2006 Aug 22. PMID 16928441
- [Background] McNamara RK, Hahn CG, Jandacek R, Rider T, Tso P, Stanford KE, Richtand NM. Selective deficits in the omega-3 fatty acid docosahexaenoic acid in the postmortem orbitofrontal cortex of patients with major depressive disorder. Biol Psychiatry. 2007 Jul 1;62(1):17-24. doi: 10.1016/j.biopsych.2006.08.026. Epub 2006 Dec 22. PMID 17188654
- [Background] McNamara RK, Jandacek R, Rider T, Tso P, Stanford KE, Hahn CG, Richtand NM. Deficits in docosahexaenoic acid and associated elevations in the metabolism of arachidonic acid and saturated fatty acids in the postmortem orbitofrontal cortex of patients with bipolar disorder. Psychiatry Res. 2008 Sep 30;160(3):285-99. doi: 10.1016/j.psychres.2007.08.021. Epub 2008 Aug 20. PMID 18715653
- [Background] Murphy BL, Stoll AL, Harris PQ, Ravichandran C, Babb SM, Carlezon WA Jr, Cohen BM. Omega-3 fatty acid treatment, with or without cytidine, fails to show therapeutic properties in bipolar disorder: a double-blind, randomized add-on clinical trial. J Clin Psychopharmacol. 2012 Oct;32(5):699-703. doi: 10.1097/JCP.0b013e318266854c. PMID 22926607
- [Background] Noaghiul S, Hibbeln JR. Cross-national comparisons of seafood consumption and rates of bipolar disorders. Am J Psychiatry. 2003 Dec;160(12):2222-7. doi: 10.1176/appi.ajp.160.12.2222. PMID 14638594
- [Background] Nemets B, Stahl Z, Belmaker RH. Addition of omega-3 fatty acid to maintenance medication treatment for recurrent unipolar depressive disorder. Am J Psychiatry. 2002 Mar;159(3):477-9. doi: 10.1176/appi.ajp.159.3.477. PMID 11870016
- [Background] Nemets H, Nemets B, Apter A, Bracha Z, Belmaker RH. Omega-3 treatment of childhood depression: a controlled, double-blind pilot study. Am J Psychiatry. 2006 Jun;163(6):1098-100. doi: 10.1176/ajp.2006.163.6.1098. PMID 16741212
- [Background] Peet M, Murphy B, Shay J, Horrobin D. Depletion of omega-3 fatty acid levels in red blood cell membranes of depressive patients. Biol Psychiatry. 1998 Mar 1;43(5):315-9. doi: 10.1016/s0006-3223(97)00206-0. PMID 9513745
- [Background] Peet M, Horrobin DF. A dose-ranging study of the effects of ethyl-eicosapentaenoate in patients with ongoing depression despite apparently adequate treatment with standard drugs. Arch Gen Psychiatry. 2002 Oct;59(10):913-9. doi: 10.1001/archpsyc.59.10.913. PMID 12365878
- [Background] Rondanelli M, Giacosa A, Opizzi A, Pelucchi C, La Vecchia C, Montorfano G, Negroni M, Berra B, Politi P, Rizzo AM. Effect of omega-3 fatty acids supplementation on depressive symptoms and on health-related quality of life in the treatment of elderly women with depression: a double-blind, placebo-controlled, randomized clinical trial. J Am Coll Nutr. 2010 Feb;29(1):55-64. doi: 10.1080/07315724.2010.10719817. PMID 20595646
- [Background] Ross BM, Seguin J, Sieswerda LE. Omega-3 fatty acids as treatments for mental illness: which disorder and which fatty acid? Lipids Health Dis. 2007 Sep 18;6:21. doi: 10.1186/1476-511X-6-21. PMID 17877810
- [Background] Simopoulos AP. Essential fatty acids in health and chronic diseases. Forum Nutr. 2003;56:67-70. No abstract available. PMID 15806801
- [Background] Stahl LA, Begg DP, Weisinger RS, Sinclair AJ. The role of omega-3 fatty acids in mood disorders. Curr Opin Investig Drugs. 2008 Jan;9(1):57-64. PMID 18183532
- [Background] Stoll AL, Severus WE, Freeman MP, Rueter S, Zboyan HA, Diamond E, Cress KK, Marangell LB. Omega 3 fatty acids in bipolar disorder: a preliminary double-blind, placebo-controlled trial. Arch Gen Psychiatry. 1999 May;56(5):407-12. doi: 10.1001/archpsyc.56.5.407. PMID 10232294
- [Background] Su KP, Huang SY, Chiu CC, Shen WW. Omega-3 fatty acids in major depressive disorder. A preliminary double-blind, placebo-controlled trial. Eur Neuropsychopharmacol. 2003 Aug;13(4):267-71. doi: 10.1016/s0924-977x(03)00032-4. PMID 12888186
- [Background] Su KP, Huang SY, Chiu TH, Huang KC, Huang CL, Chang HC, Pariante CM. Omega-3 fatty acids for major depressive disorder during pregnancy: results from a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2008 Apr;69(4):644-51. doi: 10.4088/jcp.v69n0418. PMID 18370571
- [Background] Sublette ME, Bosetti F, DeMar JC, Ma K, Bell JM, Fagin-Jones S, Russ MJ, Rapoport SI. Plasma free polyunsaturated fatty acid levels are associated with symptom severity in acute mania. Bipolar Disord. 2007 Nov;9(7):759-65. doi: 10.1111/j.1399-5618.2007.00387.x. PMID 17988367
- [Background] Sublette ME, Ellis SP, Geant AL, Mann JJ. Meta-analysis of the effects of eicosapentaenoic acid (EPA) in clinical trials in depression. J Clin Psychiatry. 2011 Dec;72(12):1577-84. doi: 10.4088/JCP.10m06634. Epub 2011 Sep 6. PMID 21939614
- [Background] Tajalizadekhoob Y, Sharifi F, Fakhrzadeh H, Mirarefin M, Ghaderpanahi M, Badamchizade Z, Azimipour S. The effect of low-dose omega 3 fatty acids on the treatment of mild to moderate depression in the elderly: a double-blind, randomized, placebo-controlled study. Eur Arch Psychiatry Clin Neurosci. 2011 Dec;261(8):539-49. doi: 10.1007/s00406-011-0191-9. Epub 2011 Feb 12. PMID 21318452
- [Background] Tanskanen A, Hibbeln JR, Hintikka J, Haatainen K, Honkalampi K, Viinamaki H. Fish consumption, depression, and suicidality in a general population. Arch Gen Psychiatry. 2001 May;58(5):512-3. doi: 10.1001/archpsyc.58.5.512. No abstract available. PMID 11343534
- [Background] Umhau JC, Zhou W, Carson RE, Rapoport SI, Polozova A, Demar J, Hussein N, Bhattacharjee AK, Ma K, Esposito G, Majchrzak S, Herscovitch P, Eckelman WC, Kurdziel KA, Salem N Jr. Imaging incorporation of circulating docosahexaenoic acid into the human brain using positron emission tomography. J Lipid Res. 2009 Jul;50(7):1259-68. doi: 10.1194/jlr.M800530-JLR200. Epub 2008 Dec 26. PMID 19112173
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] McPhilemy G, Byrne F, Waldron M, Hibbeln JR, Davis J, McDonald C, Hallahan B. A 52-week prophylactic randomised control trial of omega-3 polyunsaturated fatty acids in bipolar disorder. Bipolar Disord. 2021 Nov;23(7):697-706. doi: 10.1111/bdi.13037. Epub 2021 Jan 10. PMID 33340432